CLINICAL TRIAL: NCT04110717
Title: Electrical Vestibular Nerve Stimulation (VeNS) Together With a Lifestyle Modification Program, Compared to a Sham Control With a Lifestyle Modification Program, as a Means of Reducing Excess Body Weight and Body Fat.
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) Compared to Sham Control as a Means of Reducing Excess Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: University College Dublin (Other); Exploristics Ltd (Unknown); Compliance Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050719-UCD
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Overweight; Obesity; Overweight and Obesity; Overweight or Obesity; Metabolic Syndrome
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Device Group (Experimental): 25 subjects randomised to receive active device use plus lifestyle intervention for 3 months.
  Interventions: Device: Vestal Device; Behavioral: Hypocaloric Diet
- Control Device Group (Placebo Comparator): 25 subjects randomised to receive control device use plus lifestyle intervention for 3 months.
  Interventions: Device: Control Device; Behavioral: Hypocaloric Diet

INTERVENTIONS:
Device: Vestal Device — Vestibular nerve stimulator
  Arms: Active Device Group
Device: Control Device — Control Device
  Arms: Control Device Group
Behavioral: Hypocaloric Diet — Hypocaloric diet

SUMMARY:
A randomized, double blind sham controlled clinical trial to evaluate the efficacy of vestibular nerve stimulation (VeNS), together with a lifestyle modification program, compared to a sham control with a lifestyle modification programme, as a means of reducing excess body weight and body fat.

ELIGIBILITY:
Inclusion Criteria:

* 1. Body mass index (BMI) ≥ 25 kg/m2 2. Males or Females. Note females of child-bearing potential must have a negative urine pregnancy test They should agree to follow a physician-approved contraceptive regimen for the duration of the study period (other than DMPA injections as this causes weight gain).

  3. 18-80 years of age inclusive on starting the study. 4. Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with: trying to use the device on a daily basis; the hypocaloric diet weight loss program; and this provided weight loss support and mentoring.

  5. Agreement not to use of prescription, or over-the-counter, weight loss preparations for the duration of the trial.

  6. Agreement not to start smoking tobacco or marijuana for the duration of the study.

  7. Access to Wi-Fi (to connect iPod to internet)

Exclusion Criteria:

* 1. History of vestibular dysfunction or other inner ear disease as indicated by the screening questions.

  2. History of bariatric surgery, or gastric resection. 3. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.

  4. History of weight loss device implantation (e.g. VBloc Maestro or Abiliti). 5. Use of a non-invasive weight loss device (e.g. Modius) 6. Hypothyroidism requiring current treatment with levothyroxine (e.g. Levo-T, Synthroid, Thyroxine) (Other thyroid disorder patients on stable treatment for at least 3 months are acceptable).

  7. Other endocrinological causes of weight gain (e.g. Cushing's disease, Cushing's syndrome or acromegaly) 8. Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working).

  9. Diagnosis of cirrhosis, chronic pancreatitis, or liver, kidney or heart failure.

  10. Treatment with prescription weight-loss drug therapy in the 6 months before starting the study.

  11. Tobacco or marijuana smoking in the 6 months before starting and for the duration of the study.

  12. Known genetic cause of obesity (e.g., Prader-Willi Syndrome). 13. Body weight change of more than 20% in either direction within the previous year.

  14. Physician-prescribed diet, and/ or current, active member of an organized weight loss program.

  15. Diabetes mellitus (Types 1 & 2). 16. Diagnosis of epilepsy or use of anti-epileptic medication within six months of starting the study (e.g. for the treatment of peripheral neuropathy) 17. Chronic (more than a month of daily use) treatment with opioid analgesic drugs within the last 6 months.

  18. Regular use (more than twice a month) of anti-histamine medication within the last 6 months.

  19. Use of oral or intravenous corticosteroid medication within 6 months of starting the study.

  20. Use of the beta-blockers atenolol, metoprolol or propranolol within 3 months of starting the study.

  21. Current alterations in treatment regimens of anti-depressant medication for whatever reason (including tricyclic antidepressants) (Note: stable treatment regimen for prior 6 months acceptable).

  22. An active diagnosis of cancer. 23. A myocardial infarction within the preceding year. 24. A history of stroke or severe head injury (as defined by a head injury that required craniotomy or endotracheal intubation). (In case this damaged the neurological pathways involved in vestibular stimulation).

  25. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).

  26. Psychiatric disorders (including untreated severe depression, schizophrenia, substance abuse, eating disorder etc.) 27. Current participant in another weight loss study or other clinical trial. 28. Have a family member who is currently participating or is planning to participate in this study.

  29. Pregnancy 30. History of migraine headaches

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Total body weight loss | 12 weeks
  In kg

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No